CLINICAL TRIAL: NCT03716869
Title: Randomized Controlled Trial of Universal vs. Targeted School Screening for Adolescent Major Depressive Disorder
Brief Title: Universal vs. Targeted School Screening for Adolescent Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Deepa Sekhar, Associate Professor, Department of Pediatrics, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: STUDY00010090; R40MC31765 (Other Grant/Funding Number: Health Resources and Services Administration)
Record Dates: First submitted 2018-10-15; First posted 2018-10-23 (Actual); Results first posted 2022-03-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-04

CONDITIONS: Major Depressive Disorder; Major Depressive Episode
Keywords: adolescent; mental health; depression; suicide
MeSH Terms: conditions — Depressive Disorder, Major; Psychological Well-Being; Depression; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted Screening Arm (Current Process) (No Intervention): Students randomized to the targeted screening arm will complete their routine school-based health screenings. Students will be followed through the academic year for referrals to the Student Assistance Program (SAP). SAP currently exists in all Pennsylvania (PA) schools and functions like a triage service. If a student exhibits behavior concerning for MDD (raised by any contact, e.g. teachers, nurse, parent, peer, or even self-referral), SAP will triage the student and based on the initial assessment provide recommendations for school or community-based services.
- Universal Screening Arm (Intervention) (Experimental): Students randomized to the universal screening arm will complete the Patient Health Questionnaire (PHQ-9) during the academic year. This screening tool includes nine close-ended questions with a scoring system ranging from 0 to 27. Scores >10 are considered a "positive" screen. Students with a positive PHQ-9 result will then proceed to SAP triage as per the current process for those referred via the targeted screening arm.
  Interventions: Other: Universal Screening Arm

INTERVENTIONS:
Other: Universal Screening Arm — Students with PHQ-9 score >10, corresponding to a positive MDD screen, will proceed through the same SAP triage process as students referred by traditional means.
  SAP triage will determine MDD identification. As SAP triage is not diagnostic, MDD identification is based on SAP recommendations for MDD related school or community services.
  Treatment engagement will be tracked per current SAP processes.
  To immediately identify and address suicidal intent, the survey will flag a positive response to PHQ-9 question 9 in real time. A suicidal student would proceed directly to management through the school crisis plan.
  Students in the intervention arm will also be tracked for behavior concerning for MDD at any point in the school year prompting SAP triage referral.
  Arms: Universal Screening Arm (Intervention)

SUMMARY:
The primary goal of the proposed study is to compare the effectiveness of universal school based screening for adolescent major depressive disorder to the current school process of targeted screening based on concerning behavior.

DETAILED DESCRIPTION:
The prevalence of annual major depressive disorder (MDD) episodes has increased by greater than 50% from 2008 to 2015 among US adolescents. Paralleling the rise in MDD, suicide is now the 2nd leading cause of adolescent deaths. Despite the US Preventive Services Task Force (USPSTF) 2009 endorsement of universal screening for adolescent MDD in primary care, MDD screening occurs in less than 2% of office visits.

The primary goal of the proposed study is to compare the effectiveness of universal versus targeted adolescent MDD screening in a school setting. Universal screening was chosen to be conducted in schools because, compared to medical settings; schools are more likely to regularly engage with adolescents.

The hypothesis is that universal school-based screening with the validated Patient Health Questionnaire (PHQ) will result in increased rates of MDD screening, identification and treatment engagement. The Penn State team brings a breadth of experience in pediatrics, community-engaged research, adolescent health, psychiatry and engagement with minority populations.

ELIGIBILITY:
Inclusion Criteria:

* Students in grades 9-12 at 14 public schools in Pennsylvania. This is a change from the originally anticipated 16 schools, as 2 were unable to continue participation. Anticipated enrollment numbers will be updated once the data are finalized.

HRSA funding for primarily rural school districts (only one is urban). PCORI funding for urban school districts.

Exclusion Criteria:

* Students whose parents complete the opt-out consent
* Students not enrolled in one of the participating schools
* Students not in grades 9-12
* Students with disabilities that are deemed unable to participate by the school district

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12909 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepa Sekhar, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- The Pennsylvania State University, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data set
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data available December 2022, details of how long the data will be available are TBD
Access Criteria: At this time, data would be accessed by contacting the Principal Investigator, Deepa Sekhar.

REFERENCES:
- [Derived] Sekhar DL, Batra E, Schaefer EW, Walker-Harding LR, Pattison KL, Molinari A, Rosen P, Kraschnewski JL, Waxmonsky JG. Adolescent Suicide Risk Screening: A Secondary Analysis of the SHIELD Randomized Clinical Trial. J Pediatr. 2022 Dec;251:172-177. doi: 10.1016/j.jpeds.2022.07.036. Epub 2022 Aug 6. PMID 35944722
- [Derived] Sekhar DL, Schaefer EW, Waxmonsky JG, Walker-Harding LR, Pattison KL, Molinari A, Rosen P, Kraschnewski JL. Screening in High Schools to Identify, Evaluate, and Lower Depression Among Adolescents: A Randomized Clinical Trial. JAMA Netw Open. 2021 Nov 1;4(11):e2131836. doi: 10.1001/jamanetworkopen.2021.31836. PMID 34739064
- [Derived] Sekhar DL, Pattison KL, Confair A, Molinari A, Schaefer EW, Waxmonsky JG, Walker-Harding LR, Rosen P, Kraschnewski JL. Effectiveness of Universal School-Based Screening vs Targeted Screening for Major Depressive Disorder Among Adolescents: A Trial Protocol for the Screening in High Schools to Identify, Evaluate, and Lower Depression (SHIELD) Randomized Clinical Trial. JAMA Netw Open. 2019 Nov 1;2(11):e1914427. doi: 10.1001/jamanetworkopen.2019.14427. PMID 31675086

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Letters sent to parents or guardians before screening detailed the project and screening instrument, the Patient Health Questionnaire-9 (PHQ-9), and offered the opportunity to opt their student out of the study. Out of 13,171 students, 262 opted out.
Groups:
- Targeted Screening Arm (Current Process): Students randomized to the targeted screening arm will complete their routine school-based health screenings. Students will be followed through the academic year for referrals to the Student Assistance Program (SAP). SAP currently exists in all Pennsylvania (PA) schools and functions like a triage service. If a student exhibits behavior concerning for major depressive disorder (MDD; raised by any contact, e.g. teachers, nurse, parent, peer, or even self-referral), SAP will triage the student and based on the initial assessment provide recommendations for school or community-based services.
- Universal Screening Arm (Intervention): Students randomized to the universal screening arm will complete the Patient Health Questionnaire (PHQ-9) during the academic year. This screening tool includes nine close-ended questions with a scoring system ranging from 0 to 27. Scores >10 are considered a "positive" screen. Students with a positive PHQ-9 result will then proceed to Student Assistance Program (SAP) triage as per the current process for those referred via the targeted screening arm.
  Universal Screening Arm: Students with PHQ-9 score >10, corresponding to a positive major depressive disorder (MDD) screen, will proceed through the same SAP triage process as students referred by traditional means.
  SAP triage will determine MDD identification. As SAP triage is not diagnostic, MDD identification is based on SAP recommendations for MDD related school or community services.
  Treatment engagement will be tracked per current SAP processes.
  To immediately identify and address suicidal intent, the survey will flag a positive response to PHQ-9 question 9 in real time. A suicidal student would proceed directly to management through the school crisis plan.
  Students in the intervention arm will also be tracked for behavior concerning for MDD at any point in the school year prompting SAP triage referral.
Period: Overall Study
Arm/Group | Targeted Screening Arm (Current Process) | Universal Screening Arm (Intervention)
Started | 6436 | 6473
Completed | 6436 | 6473
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Universal Screening Arm (Intervention): Students randomized to the universal screening arm will complete the Patient Health Questionnaire (PHQ-9) during the academic year. This screening tool includes nine close-ended questions with a scoring system ranging from 0 to 27. Scores >10 are considered a "positive" screen. Students with a positive PHQ-9 result will then proceed to SAP triage as per the current process for those referred via the targeted screening arm.
  Universal Screening Arm: Students with PHQ-9 score >10, corresponding to a positive MDD screen, will proceed through the same SAP triage process as students referred by traditional means.
  SAP triage will determine MDD identification. As SAP triage is not diagnostic, MDD identification is based on SAP recommendations for MDD related school or community services.
  Treatment engagement will be tracked per current SAP processes.
  To immediately identify and address suicidal intent, the survey will flag a positive response to PHQ-9 question 9 in real time. A suicidal student would proceed directly to management through the school crisis plan.
  Students in the intervention arm will also be tracked for behavior concerning for MDD at any point in the school year prompting SAP triage referral.
- Total: Total of all reporting groups
Arm/Group | Targeted Screening Arm (Current Process) | Universal Screening Arm (Intervention) | Total
Number analyzed (Participants) | 6436 | 6473 | 12909
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 16 [15 to 17] | 16 [15 to 17] | 16 [15 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2941 | 3005 | 5946
  Male | 3495 | 3468 | 6963
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic (any race) | 1266 | 1421 | 2687
  Non-Hispanic Black | 1571 | 1320 | 2891
  Non-Hispanic White | 2857 | 2985 | 5842
  Other or multiple races | 742 | 747 | 1489
Region of Enrollment [Number; unit: participants]
  United States | 6436 | 6473 | 12909
Grade [Count of Participants; unit: Participants]
  9th | 2430 | 1531 | 3961
  10th | 1048 | 2106 | 3154
  11th | 1932 | 1051 | 2983
  12th | 1026 | 1785 | 2811
Urban/rural [Count of Participants; unit: Participants]
  Urban | 5728 | 5735 | 11463
  Rural | 708 | 738 | 1446

OUTCOME MEASURES:

1. Primary Outcome: Major Depressive Disorder (MDD) Composite: Positive Patient Health Questionnaire-9 (PHQ-9; Universal Arm) or MDD Concern Prompting Student Assistance Program (SAP) Referral, Confirmed MDD Symptoms by SAP, Engage With One SAP Recommended Service/Treatment
Description: Universal 1) Adolescents with PHQ-9 score >10 or who at any point in the year exhibit behavior concerning for MDD prompting a SAP triage request (PHQ-9 score: min 0, max 27, higher scores=greater depression symptoms), 2) Adolescents identified with MDD by SAP triage, and 3) Adolescents who successfully engage with at least one SAP recommendation.
  Prior Sept-Nov screening adjusted per school preference.
  Targeted
  1) Adolescents with behavior concerning for MDD prompting a SAP triage request, 2) Adolescents identified with MDD by SAP triage, and 3) Adolescents who successfully engage with at least one SAP recommendation
  Concern for MDD based on a primary or secondary potentially MDD related SAP "incoming referral reason"
  SAP triage is not diagnostic, so MDD identified based on recommendations for MDD related school or community services (e.g. mental health treatment services)
  HRSA funds mostly rural schools (all rural but one school) and PCORI funds urban schools
Time Frame: up to 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Targeted Screening Arm (Current Process) | Universal Screening Arm (Intervention)
Number analyzed (Participants) | 6436 | 6473
Participants | 35 | 80
Statistical Analysis 1: Comparison: Targeted Screening Arm (Current Process) vs Universal Screening Arm (Intervention); Statistical analysis was conducted using the intent-to-treat principle. Analysis for primary and secondary outcomes that compared universal to targeted screening was conducted using mixed effects logistic regression; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.07, 95% CI 2-sided [1.39 to 3.10]

2. Secondary Outcome: MDD Screen Positive/Concern: Adolescents Who Screen Positive for MDD Either by PHQ-9 (Universal Screening Arm Only) or by Concern for MDD Prompting a Request for SAP Triage
Description: Universal screening arm: Adolescents with PHQ-9 score >10 or who at any point in the year exhibit behavior concerning for MDD prompting a self or collateral request for SAP triage (PHQ-9 score: min 0, max 27, higher scores=greater depression symptoms)
  Targeted screening arm: Adolescents with behavior concerning for MDD which prompts self or collateral request for SAP triage at any point during the school year.
  Concern for MDD is based on a primary or secondary potentially MDD related SAP "incoming referral reason".
Time Frame: up to 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Targeted Screening Arm (Current Process) | Universal Screening Arm (Intervention)
Number analyzed (Participants) | 6436 | 6473
Participants | 200 | 1026
Statistical Analysis 1: Comparison: Targeted Screening Arm (Current Process) vs Universal Screening Arm (Intervention); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.92, 95% CI 2-sided [5.07 to 6.93]

3. Secondary Outcome: Suicidal Adolescent
Description: Universal screening arm: PHQ-9 positive response to question #9 re: suicidal thoughts, which requires management by the state-mandated school crisis plan or student self or collateral report of suicidal thoughts, which requires management by the state-mandated school crisis plan (source school district).
  Targeted screening arm: Student self or collateral report of suicidal thoughts, which requires management by the state-mandated school crisis plan (source school district).
  Any student suicide attempts or completed suicides shared with the school district will also be included.
Time Frame: up to 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Targeted Screening Arm (Current Process) | Universal Screening Arm (Intervention)
Number analyzed (Participants) | 6436 | 6473
Participants | 96 | 622

4. Secondary Outcome: MDD Identification: Adolescents Confirmed With MDD Symptoms in Need of Follow-up Based on Triage by the School SAP Team
Description: Universal and targeted screening arms: Adolescents who are identified as having MDD symptoms in need of follow-up based on triage by the school SAP team.
  As SAP triage is not diagnostic, MDD identified will be based on SAP recommendations for school or community services which are MDD related (e.g. mental health treatment services).
Time Frame: up to 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Targeted Screening Arm (Current Process) | Universal Screening Arm (Intervention)
Number analyzed (Participants) | 6436 | 6473
Participants | 64 | 233
Statistical Analysis 1: Comparison: Targeted Screening Arm (Current Process) vs Universal Screening Arm (Intervention); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.30, 95% CI 2-sided [2.49 to 4.38]

5. Secondary Outcome: MDD Treatment Engagement: Successful Engagement With at Least One SAP Recommendation
Description: Universal and targeted screening arms: Adolescents who successfully engage with at least one SAP recommendation. This may be fulfilled by parental report that an appointment was successfully scheduled.
Time Frame: up to 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Targeted Screening Arm (Current Process) | Universal Screening Arm (Intervention)
Number analyzed (Participants) | 6436 | 6473
Participants | 35 | 80

6. Secondary Outcome: Student School Policy Violations and Suspensions Based on School District Data
Description: data aggregate by grade level only
  schools currently track the number of student policy violations (e.g. for drug and alcohol, violence) and student suspensions
Time Frame: up to 9 months
Population: Information was obtained from one of the participating schools in the 2018-2019 school year. The following year saw the start of the COVID-19 pandemic (2019-2020). It was ultimately decided obtaining this secondary, grade level information was a lower priority compared to the primary outcome.
  Data from this one school is reported, but no further analysis was conducted.
Measure: Count of Participants; unit: Participants
Arm/Group | Targeted Screening Arm (Current Process) | Universal Screening Arm (Intervention)
Number analyzed (Participants) | 36 | 33
Participants | 3 | 1

7. Secondary Outcome: Missed School Days
Description: data aggregate by grade level only
Time Frame: up to 9 months
Population: as for outcome 6
Measure: Number; unit: absences
Units Other Than Participants: Eligible days=180 school days x #student
Arm/Group | Targeted Screening Arm (Current Process) | Universal Screening Arm (Intervention)
Number analyzed (Participants) | 36 | 33
Number analyzed (Eligible days=180 school days x #student) | 6480 | 5940
absences | 495 | 358

8. Secondary Outcome: Grade Point Average (Gpa)
Description: data aggregate by grade level only
Time Frame: up to 9 months
Population: Information was obtained from one of the participating schools in the 2018-2019 school year. The following year saw the start of the COVID-19 pandemic (2019-2020). It was ultimately decided obtaining this secondary, grade level information was a lower priority compared to the primary outcome.
  Data from this one school is reported as summed gpa by grades randomized to each arm, but no further analysis was conducted.
Measure: Number; unit: total summed gpa per grade in each arm
Units Other Than Participants: summed max gpa (4.0) per grade/arm
Arm/Group | Targeted Screening Arm (Current Process) | Universal Screening Arm (Intervention)
Number analyzed (Participants) | 36 | 33
Number analyzed (summed max gpa (4.0) per grade/arm) | 8 | 8
total summed gpa per grade in each arm | 6.2 | 5.2

9. Secondary Outcome: Grade Advancement/Graduation: This Measure Represents the Percent of Students Promoted in Each Grade for the School (Grades 9-12, School District Data)
Description: data aggregate by grade level only
  Note: The clinical trials record previously included additional secondary outcome measures for the Keystone testing and SAT/ACT testing. However, as these data were only received from one school, and these tests are only given in specific grades, reporting these outcomes would require disclosure of the number of students in specific grades at this school. This level of detail could allow specific school identification, and the variables were removed.
Time Frame: up to 9 months
Population: Information obtained from one school in the 2018-2019 school year. The following year was the COVID-19 pandemic (2019-2020). It was decided obtaining this secondary, grade level information was a lower priority versus the primary outcome.
  For this single school all students advanced to the next grade level. Cell counts are low and reporting raw numbers would allow identification of the school, so the information is provided as a percentage.
Measure: Number; unit: % of students
Arm/Group | Targeted Screening Arm (Current Process) | Universal Screening Arm (Intervention)
Number analyzed (Participants) | 36 | 33
% of students | 100 | 100

10. Other Pre Specified Outcome: Subgroup Analyses Based on School District Demographic Data
Description: Sex (Male, Female), Ethnicity, Race, Rural/Urban
Time Frame: up to 9 months
Measure: Count of Participants; unit: Participants
Groups:
- Female (Targeted Screening): Female students who were in the control arm, identification of depressive symptoms based on observable behaviors of concern.
- Female (Universal Screening): Female students who completed the PHQ-9 for identification of depressive symptoms.
- Male (Targeted Screening): Male students who were in the control arm, identification of depressive symptoms based on observable behaviors of concern.
- Male (Universal Screening): Male students who completed the PHQ-9 for identification of depressive symptoms.
- Non-Hispanic White (Targeted Screening): Non-Hispanic white students who were in the control arm, identification of depressive symptoms based on observable behaviors of concern.
- Non-Hispanic White (Universal Screening): Non-Hispanic white students who completed the PHQ-9 for identification of depressive symptoms.
- Non-Hispanic Black (Targeted Screening): Non-Hispanic Black students who were in the control arm, identification of depressive symptoms based on observable behaviors of concern.
- Non-Hispanic Black (Universal Screening): Non-Hispanic Black students who completed the PHQ-9 for identification of depressive symptoms.
- Hispanic (Targeted Screening): Hispanic students who were in the control arm, identification of depressive symptoms based on observable behaviors of concern.
- Hispanic (Universal Screening): Hispanic students who completed the PHQ-9 for identification of depressive symptoms.
- Other (Targeted Screening): Students classified as "other" for race/ethnicity who were in the control arm, identification of depressive symptoms based on observable behaviors of concern.
- Other (Universal Screening): Students classified as "other" for race/ethnicity who completed the PHQ-9 for identification of depressive symptoms.
- Urban (Targeted Screening): Urban students who were in the control arm, identification of depressive symptoms based on observable behaviors of concern.
- Urban (Universal Screening): Urban students who completed the PHQ-9 for identification of depressive symptoms
- Rural (Targeted Screening): Rural students who were in the control arm, identification of depressive symptoms based on observable behaviors of concern.
- Rural (Universal Screening): Rural students who completed the PHQ-9 for identification of depressive symptoms
Arm/Group | Female (Targeted Screening) | Female (Universal Screening) | Male (Targeted Screening) | Male (Universal Screening) | Non-Hispanic White (Targeted Screening) | Non-Hispanic White (Universal Screening) | Non-Hispanic Black (Targeted Screening) | Non-Hispanic Black (Universal Screening) | Hispanic (Targeted Screening) | Hispanic (Universal Screening) | Other (Targeted Screening) | Other (Universal Screening) | Urban (Targeted Screening) | Urban (Universal Screening) | Rural (Targeted Screening) | Rural (Universal Screening)
Number analyzed (Participants) | 2941 | 3005 | 3495 | 3468 | 2857 | 2985 | 1571 | 1320 | 1266 | 1421 | 742 | 747 | 5728 | 5735 | 708 | 738
Participants
  Initiated treatment | 20 | 52 | 15 | 28 | 27 | 42 | 6 | 13 | 2 | 16 | 0 | 9 | 28 | 69 | 7 | 11
  SAP confirmed depressive symptoms in need of follow-up | 31 | 153 | 33 | 80 | 48 | 115 | 10 | 37 | 5 | 67 | 1 | 14 | 55 | 212 | 9 | 21
  Identified via PHQ-9 or behaviors of concern | 90 | 626 | 110 | 400 | 61 | 474 | 95 | 187 | 28 | 204 | 16 | 161 | 189 | 893 | 11 | 133
Statistical Analysis 1: Comparison: Female (Targeted Screening) vs Female (Universal Screening) vs Male (Targeted Screening) vs Male (Universal Screening); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 8.42, 95% CI 2-sided [6.71 to 10.58] — Test of interaction terms from mixed-effects logistic regression for subgroup analyses. Information above is sex x rand group interaction for identification of MDD symptoms among females. For males, OR 4.05 (95% CI 3.26-5.03); Sex x rand group interaction p=0.005 for SAP confirmation of need for follow-up. Females 4.73 (3.19-7.02) Males 2.09 (1.38-3.16) Sex x rand group interaction p=0.37 for treatment initiation. OR is not reported due to p>0.05
Statistical Analysis 2: Comparison: Non-Hispanic White (Targeted Screening) vs Non-Hispanic White (Universal Screening) vs Non-Hispanic Black (Targeted Screening) vs Non-Hispanic Black (Universal Screening) vs Hispanic (Targeted Screening) vs Hispanic (Universal Screening) vs Other (Targeted Screening) vs Other (Universal Screening); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 8.65, 95% CI 2-sided [6.58 to 11.35] — Information above is for race/ethnicity x rand group interaction for identification of MDD symptoms for non-Hispanic white students. For non-Hispanic Black students OR 2.55 (95% CI 1.97-3.31), Hispanic 7.45 (4.98-11.17), other 12.41 (7.34-21.00); Race/ethnicity x rand group p=0.007 for SAP confirmation of need for follow-up. non-Hispanic white 2.24 (1.59-3.15) non-Hispanic Black 4.19 (2.03-8.65) Hispanic 10.15 (4.06-25.36) Other 12.22 (1.59-94.12) Race/ethnicity x rand group interaction p=0.15 for treatment initiation. OR is not reported due to p>0.05
Statistical Analysis 3: Comparison: Urban (Targeted Screening) vs Urban (Universal Screening) vs Rural (Targeted Screening) vs Rural (Universal Screening); Test type: Superiority; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 5.47, 95% CI 2-sided [4.65 to 6.44] — Information above is location x rand group interaction for identification of MDD symptoms among urban students. For rural students and identification of depressive symptoms OR 13.60 (95% CI 7.28-25.42); Location x rand group interaction p=0.27 for SAP confirmation of need for follow-up. OR is not reported due to p>0.05. Location x rand group interaction p=0.36 for treatment initiation. OR is not reported due to p>0.05

ADVERSE EVENTS:
Time Frame: up to 9 months following the screening (e.g. duration of the academic year during which screening was implemented)
Description: Depression screening using the Patient Healthy Questionnaire-9 was considered a low risk procedure (answering questions). However, a data safety monitoring board met regularly throughout the study to address any issues of concern.
Arm/Group | Targeted Screening Arm (Current Process) | Universal Screening Arm (Intervention)
All-Cause Mortality (participants affected / at risk) | 0/6436 | 0/6473
Serious Adverse Events (participants affected / at risk) | 0/6436 | 0/6473
Other Adverse Events (participants affected / at risk) | 0/6436 | 0/6473

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/69/NCT03716869/Prot_SAP_000.pdf